CLINICAL TRIAL: NCT02131181
Title: Incidence, Long- Term Outcome and Factor Related to Non- Cardiac Postoperative Delirium in Elderly Patients (POD-I)
Brief Title: Incidence, Long- Term Outcome and Factor Related to Non- Cardiac Postoperative Delirium in Elderly Patients
Acronym: POD-I
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Tanyong Pipanmekaporn, MD, Chiang Mai University
Other Study IDs: ANE-131366-FB
Record Dates: First submitted 2013-11-23; First posted 2014-05-06 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Postoperative Delirium
Keywords: Delirium, postoperative delirium, elderly
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Delirium: Patients with delirium and patients without delirium

SUMMARY:
The purpose of this study is to determine the incidence, long term outcome and factor related to postoperative delirium in elderly patients after non-cardiac surgery.

DETAILED DESCRIPTION:
The investigators have process of quality assurance for the study including data dictionary, data verification of case record form and site monitoring and auditing.

ELIGIBILITY:
Inclusion Criteria:

* Age >/ 60 years
* American Society of Anesthesiologists (ASA) physical status 1-3
* Undergoing scheduled surgery
* Giving an informed consent

Exclusion Criteria:

* Impaired visual and auditory disturbance
* Cannot communicate with Thai language
* Undergoing neurosurgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing scheduled non-cardiac operation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | participants will be followed for the duration of hospital stay, an expected average of 1 week.
  participants will be followed for the duration of hospital stay, an expected average of 1 week.

SECONDARY OUTCOMES:
Factor related to postoperative delirium | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Anesthetic technique, Pain score, type of operation
Long-term outcomes (cognitive impairment) | 3 and 6 months after operation
  This outcome will measure only patients who develop delirium after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Tanyong Pipanmekaporn, MD, Principal Investigator — Department of Anesthesiology, Faculty ofMedicine, Chiang Mai, University, Chiang Mai, Thailand
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Chiang Mai University, Maung, Chiang Mai, Thailand

REFERENCES:
- [Derived] Banjongrewadee M, Wongpakaran N, Wongpakaran T, Pipanmekaporn T, Punjasawadwong Y, Mueankwan S. The role of perceived stress and cognitive function on the relationship between neuroticism and depression among the elderly: a structural equation model approach. BMC Psychiatry. 2020 Jan 20;20(1):25. doi: 10.1186/s12888-020-2440-9. PMID 31959135
- See also: Faculty of Medicine, Chiang Mai, Thailand — http://WWW.med.cmu.ac.th